CLINICAL TRIAL: NCT06076785
Title: Impact of ODYSight in the Management of patientS With imparairEd Visual acuitY (ODYSSEY).
Brief Title: Impact of ODYSight in the Management of patientS With imparairEd Visual acuitY
Acronym: ODYSSEY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tilak Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: TIL-003
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Impaired Visual Acuity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OdySight users: OdySight users between 07/21/2021 and 11/14/2022 who performed Visual Acuity testing through OdySight and according to standard practice.
  Interventions: Device: OdySight

INTERVENTIONS:
Device: OdySight — At home measurements of visual acuity through a mobile app.

SUMMARY:
Previous investigations have demonstrated the agreement between OdySight® and standardised methods in the evaluation of near visual acuity. The app allows for remote monitoring of this parameter with tracking changes. In case of decrease in visual acuity, a notification is sent to both patient and ophthalmologist. The aim of this study is to evaluate the medical relevance of OdySight® features in the management of patients suffering from impaired visual acuity.

DETAILED DESCRIPTION:
Near or distance vision impairment is affecting more and more patients each year and the prevalence is about 2.2 billion people around the world. It has been estimated that in almost half of the cases, the vision impairment has not yet been addressed or could have been prevented. The most important causes of vision impairment are:

* Age-related macular degeneration (AMD),
* Cataract,
* Diabetic retinopathy,
* Glaucoma,
* Uncorrected refracted errors. Among the strategies setup to address vision impairment, preventive care and follow-up treatment and recurrent vision monitoring are the most performant. Standard clinical care requiring patient to physically attend can be a burden for an effective care.

Remote monitoring of visual acuity and follow-up of patients suffering from visual impairment using home-based solutions have known a great outbreak in the las few years. The use of smartphones and tablets supporting applications developed to monitor and evaluate patient's vision has considerably evolved. Moreover, the recent COVID-19 pandemic underlined the need to develop qualified remote care systems to enhance healthcare access.

In the last decade, several tools were developed in the field of ophthalmology for visual function self assessment. The Visual Acuity (VA) testing is the most performed ophthalmologic examination to evaluate patient's potential visual impairment and can be tested either classically with letters optotype charts and projection systems or more recently with the help of digital tools. These tools allow patients to evaluate their VA using applications designed for smartphones, tablets, or computers.

In the standard clinical practice, the VA testing is mostly performed using a Snellen chart (black letters and optotypes of different sizes printed on a white chart), developed in 1862. This tool has been progressively improved, notably with the development of ETDRS charts, considered more accurate and that are thus used in research. These tools required the patient to physically attend the clinical examination, which is sometimes difficult to achieve considering patient mobility issues (age, disability, lack of transportation…), the lack of clinical practices in some areas, or other reasons.

Digital VA testing tools are an interesting alternative to the standard tests performed in clinic.

Nevertheless, their development implies a clinical validation research and certification, to be used for patient ophthalmic care.

Several studies have proved the reliability of digital systems for VA measurement, in remotely operated systems. In 2012, the equivalence of VA measurement using a computer-based logarithmic (logMAR) chart with the standard examination in the physical presence of an optometrist was shown. There was no statistically significant difference between the median VA measurement assessed by the two methods (physical optometrist or remote computer-based system).

The feasibility and the accuracy of a smartphone-based method for VA testing has been addressed in 2014, in the context of Early Treatment for Diabetic Retinopathy Study (ETDRS) testing, using the SightBookTM application. The results of the study evidenced test-retest high reliability and concordance with EDTRS distance VA testing and standard near vision testing.

More recently, VA testing methods have been compared using standard ETDRS chart, near chart and a smartphone-based eye chart application. The study concludes in favour of an equivalent efficiency of the three methods, suggesting a potential interest for remote VA-testing especially when standard clinical examination is not possible or difficult.

Another study, evaluating a smartphone-based VA testing (logMAR) reliability for test-retest compared to standard care showed promising results for remote healthcare and accessibility.

Interestingly, remote VA testing has been shown to be efficient in both adults and children.

The COVID-19 pandemic challenged standard ophthalmologic practice and revealed an acute need of remote healthcare access that emphasizes the development of more efficient tools for VA monitoring and clinical visit scheduling when required.

OdySight® is a medical application intended for patients 18 years of age and older for self-evaluation of visual parameters: near visual acuity and symptoms such as metamorphopsia and scotoma. The test results are sent to the doctor.

OdySight® does not provide any interpretation of the test results and is not intended to provide a diagnosis. OdySight® helps patients to determine whether they need to consult a doctor for diagnosis and treatment.

Three clinical studies have been conducted to evaluate the Odysight® application efficiency compared to standard ophthalmologic care.

In 2019, a prospective, open-labelled, single-arm, single-site study has been performed to compare the results of gold standard VA testing (Sloan ETDRS letter chart for near and distance vision testing), contrast sensitivity (Pelli-Robson chart), and metamorphopsia/scotoma (Amster Grid). The analysis showed a concordance between the results obtained with the OdySight® VA module and the Sloan ETDRS (near and distance). No significant difference has been shown between the OdySight® Amsler Grid module and standard metamorphopsia/scotoma testing. On the other hand, a broader disagreement has been pointed out for the evaluation of contrast sensitivity between the standard Pelli-Robson test and the OdySight® module, which would require more investigation.

The overall results are in favour of using the OdySight® application for remote monitoring of vision between clinic visits and potential assistance for follow-up scheduling.

In 2021, the implementation and clinical efficacy of the OdySight® application was evaluated in a study involving patients (n=60) with oedematous maculopathies receiving standard care. Patients were offered to use OdySight® to self-evaluate changes in their VA. The use of the application and the processing of notifications for VA decrease by the clinical team was analysed for one year to assess the feasibility and the reliability of the system. In all, about 60% of the patients completed at least one test following the prescription and almost 25% of the patients were still using the application after one month. During this trial, 19 notifications for VA decrease were processed by the clinical team in an average of less than 6 days. The decrease in VA was detected with a sensitivity of 92% and a specificity of 99%.

An observational, retrospective, multicentric study, published in 2022, was conducted to evaluate the additional value of using the OdySight® application in addition to a standard follow-up for the detection of exudatives recurrences in patients suffering from macular oedema. In all, 123 patients (149 eyes) were included in the study. The sensitivity of the alerts for the detection of recurrences was around 30%, and the specificity reached 84%. In total, 12 alerts on 39 detected a recurrence and 8 of them resulted in rescheduling or advancement of intravitreal injection. Although the sensitivity and the specificity appear to be a bit low, exudatives recurrences not being necessarily associated to a decrease in VA, the results of the study confirm that OdySight® use can be of interest in the detection of recurrence in advance and allow an anticipated readjustment of the treatment in addition with a standard care follow-up.

ELIGIBILITY:
Inclusion Criteria:

* OdySight® user (between 07/21/2021 and 11/14/2022),
* Performed at least 3 tests on the same eye (minimum number of tests to trigger an alert).

Exclusion Criteria:

* Opposition to personal data collection and processing,
* Patient's death is documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with a near visual acuity between 0.0 and 1.0 logMAR in at least one eye, and binocular VA equal to or better than 0.5 logMAR are targeted for this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Impact of OdySight® in the management of patients suffering from impaired visual acuity. | At least 3 months of follow-up.
  Number of patients concerned by one or more OdySight® notification(s) for visual acuity decrease followed by a visit where at least one of the following situations is noticed:
  * Visual acuity decrease
  * Anatomic ophthalmic deterioration
  * Prescription impact
  * Second eye newly affected and/or development of the pathology to the second eye

SECONDARY OUTCOMES:
Performances of OdySight® in tracking visual acuity decrease and/or anatomic change. | At least 3 months of follow-up.
  Sensitivity, specificity, Positive Predicted Value and Negative Predicted Value of OdySight® in tracking visual acuity decrease and/or anatomic change with subgroups analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte BROUSSEAU, MD, Principal Investigator — Centre Ophtalmologique Ophtalliance; Maddalena QUARANTA, MD, Principal Investigator — Centre Ophtalmologique Rabelais; Vincent GUALINO, MD, Principal Investigator — Clinique Honoré Cave; Jean-François GIRMENS, MD, Principal Investigator — Hopital des XV-XX; Isabelle FOURNIER, MD, Principal Investigator — Institut ophtalmologique Sourdille Atlantique; Marie-Noëlle GUILLEMOT, MD, Principal Investigator — Institut ophtalmologique Sourdille Atlantique; Jean-François BOULET, MD, Principal Investigator — Cabinet d'ophtalmologie; Pierre-Olivier LAFONTAINE, MD, Principal Investigator — Centre Ophtalmologique Oculus; Joël UZZAN, MD, Principal Investigator — Clinique Mathilde; Viviane VINH, MD, Principal Investigator — Centre d'Ophtalmologie du Dauphiné
Locations (8):
- France (8):
  - Centre Ophtalmologique Oculus, Chambéry, Auvergne-Rhône-Alpes
  - Centre Ophtalmologique Rabelais, Lyon, Auvergne-Rhône-Alpes
  - SELARL Dr Boulet, Évreux, Normandy
  - Clinique Mathilde, Rouen, Normandy
  - Clinique Honoré Cave, Montauban, Occitanie
  - Institut Ophtalmologique de l'Ouest Jules Verne, Nantes, Pays de la Loire Region
  - Institut ophtalmologique Sourdille Atlantique, Saint-Herblain, Pays de la Loire Region
  - Hôpital des XV-XX, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Causes of blindness and vision impairment in 2020 and trends over 30 years, and prevalence of avoidable blindness in relation to VISION 2020: the Right to Sight: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e144-e160. doi: 10.1016/S2214-109X(20)30489-7. Epub 2020 Dec 1. PMID 33275949
- [Background] Claessens JLJ, Geuvers JR, Imhof SM, Wisse RPL. Digital Tools for the Self-Assessment of Visual Acuity: A Systematic Review. Ophthalmol Ther. 2021 Dec;10(4):715-730. doi: 10.1007/s40123-021-00360-3. Epub 2021 Jun 25. PMID 34169468
- [Background] Srinivasan K, Ramesh SV, Babu N, Sanker N, Ray A, Karuna SM. Efficacy of a remote based computerised visual acuity measurement. Br J Ophthalmol. 2012 Jul;96(7):987-90. doi: 10.1136/bjophthalmol-2012-301751. Epub 2012 Apr 26. PMID 22539747
- [Background] Yeung WK, Dawes P, Pye A, Neil M, Aslam T, Dickinson C, Leroi I. eHealth tools for the self-testing of visual acuity: a scoping review. NPJ Digit Med. 2019 Aug 22;2:82. doi: 10.1038/s41746-019-0154-5. eCollection 2019. PMID 31453377
- [Background] Williams AM, Kalra G, Commiskey PW, Bowers EMR, Rudolph BR, Pitcher MD, Dansingani KK, Jhanji V, Nischal KK, Sahel JA, Waxman EL, Fu R. Ophthalmology Practice During the Coronavirus Disease 2019 Pandemic: The University of Pittsburgh Experience in Promoting Clinic Safety and Embracing Video Visits. Ophthalmol Ther. 2020 Sep;9(3):1-9. doi: 10.1007/s40123-020-00255-9. Epub 2020 May 6. PMID 32377502
- [Background] Tiraset N, Poonyathalang A, Padungkiatsagul T, Deeyai M, Vichitkunakorn P, Vanikieti K. Comparison of Visual Acuity Measurement Using Three Methods: Standard ETDRS Chart, Near Chart and a Smartphone-Based Eye Chart Application. Clin Ophthalmol. 2021 Feb 26;15:859-869. doi: 10.2147/OPTH.S304272. eCollection 2021. PMID 33664563
- [Background] Miller JM, Jang HS, Ramesh D, Gonzalez Marshall MS, Yescas S, Harvey EM. Telemedicine distance and near visual acuity tests for adults and children. J AAPOS. 2020 Aug;24(4):235-236. doi: 10.1016/j.jaapos.2020.06.003. Epub 2020 Jul 30. PMID 32739362
- [Background] Iskander M, Hu G, Sood S, Heilenbach N, Sanchez V, Ogunsola T, Chen D, Elgin C, Patel V, Wronka A, Al-Aswad LA. Validation of the New York University Langone Eye Test Application, a Smartphone-Based Visual Acuity Test. Ophthalmol Sci. 2022 Jun 15;2(3):100182. doi: 10.1016/j.xops.2022.100182. eCollection 2022 Sep. PMID 36245756
- [Background] Kielwasser G, Kodjikian L, Dot C, Burillon C, Denis P, Mathis T. Real-Life Value of the Odysight(R) Application in At-Home Screening for Exudative Recurrence of Macular Edema. J Clin Med. 2022 Aug 26;11(17):5010. doi: 10.3390/jcm11175010. PMID 36078941
- [Background] Guigou S, Michel T, Merite PY, Coupier L, Meyer F. Home vision monitoring in patients with maculopathy: Real-life study of the OdySight application. J Fr Ophtalmol. 2021 Jun;44(6):873-881. doi: 10.1016/j.jfo.2020.09.034. Epub 2021 May 20. PMID 34024655
- [Background] Brucker J, Bhatia V, Sahel JA, Girmens JF, Mohand-Said S. Odysight: A Mobile Medical Application Designed for Remote Monitoring-A Prospective Study Comparison with Standard Clinical Eye Tests. Ophthalmol Ther. 2019 Sep;8(3):461-476. doi: 10.1007/s40123-019-0203-9. Epub 2019 Jul 25. PMID 31346977
- [Background] Allen L, Thirunavukarasu AJ, Podgorski S, Mullinger D. Novel web application for self-assessment of distance visual acuity to support remote consultation: a real-world validation study in children. BMJ Open Ophthalmol. 2021 Sep 30;6(1):e000801. doi: 10.1136/bmjophth-2021-000801. eCollection 2021. PMID 34651083